CLINICAL TRIAL: NCT00810680
Title: Use of Valproic Acid in Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Study of Efficacy and Safety of Valproic Acid in Chronic Lymphocytic Leukemia (CLL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr. Vinod Raina, Institute Rotary Cancer Hospital, AIIMS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCH-VAL-01
Record Dates: First submitted 2008-10-21; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; relapsed; refractory; valproic acid; valproate
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valproic acid (Experimental)
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Valproic acid — Tab. Valproic acid will be started at a dose of 10 mg per kg per day in two or three divided doses. If well tolerated the dose will be increased to a maximum of 20 mg per kg per day and continued for a period of 3 months. The drug will be continued for another 3 months for a maximum of 6 months in responding patients. The drug will be stopped in all those who develop intolerable side effects or develop disease progression during therapy.
  Other Names: Valproate; Sodium Valproate; Depakote

SUMMARY:
The purpose of this study is to determine whether Valproic acid, as a single agent is effective in the treatment of Chronic Lymphocytic Leukemia which has relapsed or is refractory to therapy with standard drugs.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is a disease characterized by a prolonged clinical course. Though various drugs such as alkylating agents, antimetabolites such as fludarabine and targeted antibodies such as rituximab are effective against this condition, relapses are frequent and cure is rare. There exists a subset of CLL patients who are refractory to many of these first line agents. Though one or the other of the above mentioned class of drugs can be substituted for patients who have relapsed or have refractory disease, no therapy has been conclusively proven to have survival advantage in this condition. The costs and toxicities add to the burden of these therapies. Valproic acid is a well studied drug used for the treatment of epilepsy for over 30 years. It has a well documented side effect profile, is generally well tolerated and is inexpensive. Recently, it has been shown to be an inhibitor of the enzyme, Histone de-acetylase(HDAC). Inhibition of HDAC promotes apoptosis, and could lead to the death of CLL cells which harbor defective apoptotic mechanisms. In vitro studies have proven the ability of therapeutic concentrations of Valproic acid to achieve cell kill in cultures of CLL cells. This study aims to identify whether valproic acid, used in standard doses has single agent activity against CLL and to assess its tolerance in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Active CLL (as defined by the National Cancer Institute Working Group)
* Patients must have received at least one prior therapy for CLL and have been treated with a nucleoside analogue.
* Age 18 years or older.
* Good general condition as defined by an Eastern cooperative oncology group- performance status (ECOG-PS) </=2.
* Absolute neutrophil count>1500/cmm and platelet count >30,000/cmm unless the low counts are due to the disease.
* Adequate liver function (bilirubin<2 mg/dL,ASTorALT <3Xthe upper limit of normal) and renal function (serum creatinine<2 mg/dL or creatinine clearance>30 mL/min) unless abnormalities are as a result of disease involvement.
* Full recovery from previous treatments.

Exclusion Criteria:

* Any therapy for CLL within 4 weeks before initiating treatment on this study.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Best clinical response as defined by NCIWG criteria for CLL | 3 months

SECONDARY OUTCOMES:
Hematological toxicity (graded according to NCIWG criteria for CLL) | 3 months
Non- hematological toxicity (graded according to NCI common toxicity criteria) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Raina, MD, FRCP, Principal Investigator — Institute Rotary Cancer Hospital, AIIMS, New delhi, India
Locations (1):
- Institute Rotary Cancer Hospital, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Bokelmann I, Mahlknecht U. Valproic acid sensitizes chronic lymphocytic leukemia cells to apoptosis and restores the balance between pro- and antiapoptotic proteins. Mol Med. 2008 Jan-Feb;14(1-2):20-7. doi: 10.2119/2007-00084.Bokelmann. PMID 17973028